CLINICAL TRIAL: NCT04911660
Title: Randomized, Double-blind, Placebo-controlled Crossover Trial Assessing the Impact of the SGLT2 Inhibitor Empagliflozin on Urinary Supersaturations in Kidney Stone Formers
Brief Title: Impact of the SGLT2 Inhibitor Empagliflozin on Urinary Supersaturations in Kidney Stone Formers
Acronym: SWEETSTONE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Boehringer Ingelheim (Industry); University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2020-02679
Record Dates: First submitted 2021-05-06; First posted 2021-06-03 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Kidney Stone
Keywords: Kidney stones; Empagliflozin; Supersaturation
MeSH Terms: conditions — Kidney Calculi | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Eligible individuals will be randomized in equal proportions to 25 mg empagliflozin or placebo, taken once daily per os in the morning. Placebo will be administered to individuals randomized to that treatment in a form identical to empagliflozin. Patients will remain on the assigned IMP for 14 days. The following 14 days (days 15 - 28) will be a wash out period without IMP intake; this wash out time can be extended to up to 6 weeks if necessary. On day 29 of the study (or later according to the length of the wash out phase), a second 14 days period with IMP intake starts (empagliflozin or placebo, whichever was not received initially).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Empagliflozin and placebo will be provided in identically looking bottles. Besides the consecutive number, packs and pack content will look identical. Therefore, all trial personnel that is involved in recruitment and care of patients, trial assessment, monitoring and analyses will be blinded to the assigned trial arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin + Placebo (Active Comparator): 1 capsule containing 25 mg empagliflozin per day for 14 days, followed by a 14-42 days wash-out phase and a second treatment phase with 1 capsule containing placebo for 14 days.
  Interventions: Drug: Empagliflozin 25 MG; Other: Placebo
- Placebo + Empagliflozin (Placebo Comparator): 1 capsule containing placebo per day for 14 days, followed by a 14-42 days wash-out phase and a second treatment phase with 1 capsule containing 25 mg empagliflozin for 14 days.
  Interventions: Drug: Empagliflozin 25 MG; Other: Placebo

INTERVENTIONS:
Drug: Empagliflozin 25 MG — 1 empagliflozin 25 mg capsule per day for 14 days
Other: Placebo — 1 placebo capsule per day for 14 days

SUMMARY:
The aim of this study is to test the effect of a new drug on the composition of the urine in kidney stone patients. This new drug (Jardiance®, substance: empagliflozin) is currently approved in Switzerland for the treatment of patients with diabetes. Data from previous studies with and without diabetes suggest that it may have a beneficial effect on the composition of the urine and thereby reduce the risk of developing kidney stones.

DETAILED DESCRIPTION:
Kidney stones - a global epidemic associated with obesity and diabetes

Kidney stones are a worldwide healthcare problem with a current lifetime risk of ~18.8 % in men and ~9.4 % in women in Western civilizations. Recurrence rates are high, up to 40 % and 75 % at 5 and 10 years, respectively. Hospitalizations, surgery and lost work time associated with kidney stones cause enormous healthcare-related expenditures. Although kidney stone disease is traditionally considered an isolated renal disorder, there is overwhelming evidence that it is in fact a systemic disease. Arterial hypertension, obesity, diabetes mellitus, gouty diathesis, dyslipidemia, cardiovascular disease, chronic kidney disease and low bone mass are much more prevalent in kidney stone formers than in non-stone formers. It is currently unknown if stone disease is a cause of this co-morbidity per se or if it is a consequence of the same underlying conditions that lead to these disorders and kidney stones. Clearly, however, these co-morbidities contribute significantly to stone-related morbidity and mortality.

The strong, positive and independent association of Body Mass Index (BMI) with kidney stone disease is well established. The magnitude of the increased risk is larger in women than in men. In addition to BMI, significant weight gain is also associated with a greater risk of developing symptomatic kidney stone disease in the future. In recent decades, the prevalence of both kidney stone disease and obesity increased significantly, irrespective of age, sex and race. In large cross-sectional analyses, the prevalence of both symptomatic and asymptomatic kidney stones increased proportionally with the number of metabolic syndrome features present. Both calcium and uric acid stones are associated with obesity, but the ratio of calcium stones to uric acid stones is lower in obese compared to non-obese stone formers, suggesting a disproportionate increase of uric acid stone disease in obesity. Absolute urinary excretion rates of stone formation promoters (calcium, phosphate, oxalate and uric acid) as well as urinary supersaturation ratios for calcium oxalate and uric acid are increased in obese individuals. In addition, there is a well documented negative association of BMI with urinary pH in both stone formers and non-stone formers, and low urinary pH is the main driver of uric acid stone formation. The latter may be explained by insulin resistance which affects the generation of renal ammonium by direct and indirect mechanisms. In contrast to urinary pH, urinary calcium excretion (the main driver for calcium stone formation) is not independently associated with BMI but rather due to other factors known to affect urinary calcium excretion (e.g. secondary to increased sodium and animal protein intake).

Supersaturation - driver of kidney stone formation

Supersaturation, the presence of a material in solution at a concentration above its own solubility, is the driving force for crystallization and therefore kidney stone formation. Relevant supersaturations for kidney stones disease in humans include calcium oxalate, brushite (calcium phosphate) and uric acid. At a supersaturation <1, crystals dissolve, at a supersaturation >1, crystals form. Urinary supersaturations calculated from ambulatory 24 h urine collections accurately reflect the long-term average supersaturation values in the urine and are highly correlated with the kidney stone composition encountered in the individual kidney stone former. Treatments that reduced stone events in Randomized Controlled Trials (RCTs) are highly correlated with reductions in urinary supersaturations. A recent analysis of a large 5-year kidney stone RCT revealed that as early as 1 week after randomization, every 10 % reduction of urinary calcium oxalate supersaturation from baseline was associated with an 8 % reduction in the risk of stone recurrence during follow-up.

SGLT2 inhibitors - a promising new drug class for kidney stone formers

Inhibitors of the sodium/glucose co-transporter isoform 2 (SLC5A2 or SGLT2) belong to a new class of oral hypoglycemic drugs. SGLT2 resides in the brush border membrane of proximal tubular cells in the kidney and reabsorbs ~90 % of glucose filtered at the glomerulus. SGLT2 inhibitors block the physiological glucose reabsorption in the proximal tubule from the glomerular filtrate, thereby inducing significant glucosuria accompanied by a reduction of blood glucose levels. Empagliflozin, the clinically best characterized SGLT2 inhibitor to date, decreases cardiovascular mortality, death from any cause, hospitalizations for heart failure, decline of GFR and need for renal replacement therapy in patients with type 2 diabetes. Some of these findings were also observed with two other SGLT2 inhibitors canagliflozin and dapagliflozin in large outcome trials. Due to their unique mode of action, SGLT2 inhibitors induce weight loss, decrease blood pressure and increase urinary volume, the latter being a very effective measure to reduce stone recurrence. Driven by promising results in RCTs, SGLT2 inhibitors are currently widely tested in non-diabetics e.g. for the treatment of heart failure, non-diabetic kidney disease, arterial hypertension or obesity (www.clinicaltrials.gov). The pleiotropic beneficial effects make SGLT2 inhibitors also a very attractive class of drugs for kidney stone formers, which often suffer concomitantly from arterial hypertension, CKD, obesity and diabetes.

Effect of SGLT2 inhibitors on bone fractures, mineral metabolism and kidney stone events

Therapy with SGLT2 inhibitors as monotherapy or add-on therapy to various glucose-lowering agents is generally well tolerated. An increased incidence of genital infections and (although rare) euglycemic ketoacidosis are known side effects of this new class of medications. The latter is mainly observed in type I diabetics and less frequently in type II diabetics. To the best of our knowledge, no cases of euglycemic ketoacidosis in individuals without diabetes treated with SGLT2 inhibitors have been reported.

In the large canagliflozin outcome study CANVAS, an increased incidence of lower extremity amputations was noted. This adverse effect has not been reported with other SGLT2 inhibitors. In addition, both canagliflozin and dapagliflozin have been associated with an increased risk of bone fractures compared to placebo. In a short term study in healthy volunteers, canagliflozin increased serum phosphate, plasma fibroblast growth factor 23 (FGF23) and plasma parathyroid hormone (PTH) and decreased the level of 1,25-dihydroxyvitamin D. Similar results were obtained in individuals with diabetes treated with dapagliflozin. In contrast, pooled analyses of phase I, II and III trials of patients with type 2 diabetes treated with empagliflozin encompassing > 15'000 patient-years of exposure did not reveal an increased rate of bone fractures, alterations of blood electrolytes, PTH, 25-dihydroxyvitamin D or bone turnover markers.

While blood electrolyte and mineral metabolism parameters in patients treated with SGLT2 inhibitors have been well studied in healthy volunteers and patients with diabetes, there is a lack of data on the impact of SGLT2 inhibition on urinary parameters, especially on parameters that influence the kidney stone formation rate. Also, to our knowledge, no studies have been conducted thus far with SGLT2 inhibitors in kidney stone formers.

Interestingly, in pooled analyses of phase I, II and III trials, the rate of kidney stone events tended to be 30-50 % lower in patients treated with 10 or 25 mg empagliflozin versus placebo. However, detailed analyses for kidney stone events in empagliflozin outcome trials have not been reported. Reported stone event rates in these pooled empagliflozin trials (0.5 - 1/100 person years) are similar to what has been observed in individuals with diabetes in three large prospective US cohorts (Nurses' Health Study I, the Nurses' Health Study II and the Health Professionals Follow-up Study. In contrast, stone event rates are considerably (10 - 100-fold) higher in patients with a history of kidney stone disease. RCTs testing dietary or pharmacologic measures for recurrence prevention typically included patients with stone event rates between 20 and 200 events/100 person-years.

In summary, SGLT2 inhibitors represent a promising new drug class for kidney stone formers. Kidney stone formers are likely to profit from the metabolic and cardiovascular effects of SGLT2 inhibition. In addition, SGLT2 inhibitors may decrease the stone formation rate. Based on the overall experience thus far, empagliflozin seems to have by far the most favorable side effect profile. Clearly, there is a dire need for clinical studies with SGLT2 inhibitors in kidney stone formers.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Age between 18 and 74 years old
* One or more kidney stone event(s) in the past
* Any past kidney stone containing ≥ 80 % of calcium or ≥ 80 % of uric acid
* HbA1c < 6.5 %

Exclusion Criteria:

* Patients with secondary causes of recurrent nephrolithiasis:
* Severe eating disorders (anorexia or bulimia)
* Chronic bowel disease, past intestinal or bariatric surgery
* Sarcoidosis
* Primary hyperparathyroidism
* Complete distal tubular acidosis
* Patients with the following medications:
* Anti-diabetic treatment (insulin and non-insulin agents)
* Patients not able or not willing to stop the following medication during the period of participation in the trial (including a time window of 4 weeks wash out prior to randomization):
* Diuretics (thiazide and loop diuretics)
* Carbonic anhydrase inhibitors (including topiramate)
* Xanthine oxidase inhibitors
* Alkali, including potassium citrate or sodium bicarbonate
* Treatment with 1,25-OH Vitamin D (calcitriol)
* Calcium supplementation
* Bisphosphonates, Denosumab, Teriparatide
* Glucocorticoids
* Obstructive uropathy, if not treated successfully
* Genito-urinary infection, if not treated successfully
* Chronic kidney disease (defined as CKD-EPI eGFR < 60 mL/min per 1.73 m2 body surface area)
* Kidney transplant
* Pregnant and lactating women [urine pregnancy test to be performed for women of childbearing potential (defined as women who are not surgically sterilized/ hysterectomized, and/ or who are postmenopausal for less than 12 months)] or women of childbearing potential that refuse to use an effective contraceptive method (birth control pill or IUD).
* Inability to understand and follow the protocol
* Known allergy to the study drug
* Participation in another interventional clinical trial within 4 weeks prior to baseline and during the current trial

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Primary outcome component 1 - calcium oxalate supersaturation in urine (empagliflozin treatment) | Oxalate supersaturation will be determined at baseline and after 14 days treatment with empagliflozin
  The primary endpoint is composed of three primary outcomes that will be assessed separately.
  1) change in calcium oxalate supersaturation after empagliflozin treatment
  Calcium oxalate supersaturation will be calculated by the Equil-2 program from the oxalate concentration in urine.
Primary outcome component 1 - calcium oxalate supersaturation in urine (placebo treatment) | Oxalate supersaturation will be determined at baseline and after 14 days treatment with placebo
  The primary endpoint is composed of three primary outcomes that will be assessed separately.
  1) change in calcium oxalate supersaturation after placebo treatment as a comparator for empagliflozin treatment
  Calcium oxalate supersaturation will be calculated by the Equil-2 program from the oxalate concentration in urine.
Primary outcome component 2 - calcium phosphate supersaturation in urine (empagliflozin treatment) | Calcium phosphate supersaturation will be determined at baseline and after 14 days treatment with empagliflozin
  The primary endpoint is composed of three primary outcomes that will be assessed separately.
  2) change in calcium phosphate supersaturation after empagliflozin treatment
  Calcium phosphate supersaturation will be calculated by the Equil-2 program from the calcium phosphate concentration in urine.
Primary outcome component 2 - calcium phosphate supersaturation in urine (placebo treatment) | Calcium phosphate supersaturation will be determined at baseline and after 14 days treatment with placebo
  The primary endpoint is composed of three primary outcomes that will be assessed separately.
  2) change in calcium phosphate supersaturation after placebo treatment as a comparator for empagliflozin treatment
  Calcium phosphate supersaturation will be calculated by the Equil-2 program from the calcium phosphate concentration in urine.
Primary outcome component 3 - uric acid supersaturation in urine (empagliflozin treatment) | Uric acid supersaturation will be determined at baseline and after 14 days treatment with empagliflozin
  The primary endpoint is composed of three primary outcomes that will be assessed separately.
  3) change in uric acid supersaturation after empagliflozin treatment
  Uric acid supersaturation will be calculated by the Equil-2 program from the uric acid concentration in urine.
Primary outcome component 3 - uric acid supersaturation in urine (placebo treatment) | Uric acid supersaturation will be determined at baseline and after 14 days treatment with placebo
  The primary endpoint is composed of three primary outcomes that will be assessed separately.
  3) change in uric acid supersaturation after placebo treatment as a comparator for empagliflozin treatment
  Uric acid supersaturation will be calculated by the Equil-2 program from the uric acid concentration in urine.

SECONDARY OUTCOMES:
Blood sodium level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Sodium level measured in mmol/l
Blood potassium level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Potassium level measured in mmol/l
Blood chloride level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Chloride level measured in mmol/l
Blood total calcium level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Total calcium level measured in mmol/l
Blood ionized calcium level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Ionized calcium level measured in mmol/l
Blood phosphate level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Phosphate level measured in mmol/l
Blood magnesium level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Magnesium level measured in mmol/l
Venous bicarbonate level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Venous bicarbonate level measured in mmol/l
Blood glucose level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Blood glucose level measured in mmol/l
Blood urea level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Urea level measured in mmol/l
Blood total cholesterol level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Total cholesterol level measured in mmol/l
Blood HDL cholesterol level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  HDL cholesterol level measured in mmol/l
Blood LDL cholesterol level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  LDL cholesterol level measured in mmol/l
Blood triglycerides level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Triglycerides level measured in mmol/l
Blood osmolality change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Osmolality measured in mmol/l
Blood creatinine level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Creatinine level measured in μmol/l
Blood uric acid level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Uric acid level measured in μmol/l
Blood 25-OH vitamine D level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  25-OH vitamine D level measured in nmol/l
Blood 1,25-OH vitamine D level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  1,25-OH vitamine D level measured in pmol/l
Venous pCO2 change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Venous pCO2 measured in mmHg
Venous pH change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Venous pH measured in pH units
Blood albumin level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Albumin level measured in g/l
Blood parathormone level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Parathormone level measured in pg/ml
Blood FGF23 level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  FGF23 level measured in pg/ml
Blood alcaline phosphatase activity change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Alcaline phosphatase activity level measured in U/l
Blood TSH activity change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  TSH activity level measured in mU/l
Blood haemoglobin A1c level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Haemoglobin A1c activity level measured in mU/l
Urine sodium level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Urine sodium level measured in mmol/l
Urine potassium level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Urine potassium level measured in mmol/l
Urine chloride level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Chloride level measured in mmol/l
Urine calcium level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Calcium level measured in mmol/l
Urine phosphate level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Phosphate level measured in mmol/l
Urine magnesium level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Magnesium level measured in mmol/l
Urine glucose level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Glucose level measured in mmol/l
Urine urea level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Urea level measured in mmol/l
Urine osmolality level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Osmolality level measured in mmol/l
Urine citrate level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Citrate level measured in mmol/l
Urine sulfate level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Sulfate level measured in mmol/l
Urine oxalate level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Oxalate level measured in μmol/l
Urine ammonia level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Ammonia level measured in μmol/l
Urine creatinine level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Creatinine level measured in μmol/l
Urine uric acid level change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Uric acid level measured in μmol/l
Urine pH change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  pH measured in pH units
Urine pCO2 change from baseline | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  pCO2 measured in mmHg
Calculated outcomes 1: estimated glomerular filtration rate (eGFR) (Blood) | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  eGFR will be derived from the serum creatinine concentration, age and sex using the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) equation
Calculated outcomes 2: titratable acid (urine) | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Titratable acid will be calculated in g/100 ml with the Equil-2 program.
Calculated outcomes 3: bicarbonate (urine) | Data collected at baseline, after 1st 14 days treatment and after 2nd 14 days treatment expected to be 6-10 weeks from baseline.
  Urine bicarbonate in mmol/l will be calculated with the Henderson-Hasselbalch equation using urine pH and urine pCO2
  HCO-3= 0.0309 x pCO2 x 10pH-6.1

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Fuster, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Inselspital, Department of Nephrology and Hypertension, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anderegg MA, Schietzel S, Bargagli M, Bally L, Faller N, Moor MB, Cereghetti GM, Roumet M, Trelle S, Fuster DG. Empagliflozin in nondiabetic individuals with calcium and uric acid kidney stones: a randomized phase 2 trial. Nat Med. 2025 Jan;31(1):286-293. doi: 10.1038/s41591-024-03330-x. Epub 2025 Jan 2. PMID 39747681
- [Derived] Schietzel S, Bally L, Cereghetti G, Faller N, Moor MB, Vogt B, Rintelen F, Trelle S, Fuster D. Impact of the SGLT2 inhibitor empagliflozin on urinary supersaturations in kidney stone formers (SWEETSTONE trial): protocol for a randomised, double-blind, placebo-controlled cross-over trial. BMJ Open. 2022 Mar 14;12(3):e059073. doi: 10.1136/bmjopen-2021-059073. PMID 35288397